CLINICAL TRIAL: NCT01850303
Title: Phase III Study Comparing Maintenance With Pemetrexed or Gemcitabine to a Surveillance in Elderly Patients (70 Years Old and More) With a Advanced Non Small Cell Lung Cancer Controlled by Induction Chemotherapy.
Brief Title: Maintenance After Induction Chemotherapy in Elderly Patients With Advanced Non-small Cell Lung Cancer
Acronym: MODEL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Intergroupe Francophone de Cancerologie Thoracique (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IFCT-1201
Record Dates: First submitted 2013-04-29; First posted 2013-05-09 (Estimated); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Non Small Cell Lung Cancer (Squamous or Non Squamous)
Keywords: Elderly; lung cancer; switch; maintenance; Elderly patients (between 70 and 89 years); NSCLC; IFCT
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Pemetrexed; Gemcitabine; Induction Chemotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Surveillance (Other)
  Interventions: Drug: Induction chemotherapy
- Maintenance (Experimental): Pemetrexed for non squamous NSCLC Gemcitabine for squamous NSCLC
  Interventions: Drug: Pemetrexed; Drug: Gemcitabine; Drug: Induction chemotherapy

INTERVENTIONS:
Drug: Pemetrexed
  Arms: Maintenance
Drug: Gemcitabine
  Arms: Maintenance
Drug: Induction chemotherapy — 4 cycles of carboplatin-paclitaxel

SUMMARY:
For elderly patient, the treatment of Non Small Cell Lung Cancer was based on monotherapy but IFCT-0501 trial begun in 2006, demonstrated that a bitherapy (carboplatin and paclitaxel) is better than monotherapy in term of overall survival and progression free survival. The current recommendations are now to administer a carboplatin based bitherapy (4 or 6 cycles). After the treatment is stopped until progression and initiation of a second line treatment. The risk of this strategy is to be confronted to a rapid disease progression during the free interval. Indeed, about 1/3 of the patients whose disease was controlled after the chemotherapy do not receive 2nd line. The concept of maintenance is based on a continuous therapeutic pressure in order to preserve the therapeutic profit obtained by the treatment of 1st line (induction chemotherapy).

There is two types of maintenance :

* continuous maintenance therapy which consists in continuing the treatment initially associated with platinum until disease progression.
* switch maintenance which consists in introducing a new treatment after the end of induction chemotherapy The two types are validated by several trials. The marketing authorization of pemetrexed was enlarged to maintenance for non squamous carcinoma.

Gemcitabine has a good tolerance profile which make possible the use in a maintenance strategy. Several trials evaluated maintenance with this product and some show benefits in term of progression free survival.

The objective of this trial is to evaluate the switch maintenance in elderly patient with a controlled disease after 4 cycles of chemotherapy carboplatin-paclitaxel.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically documented Non Small Cell Lung Cancer non resectable or non irradiable stage III or stage IV
* EGFR wild type or non feasible EGFR
* 90 >Age ≥ 70
* ECOG Performance status : 0, 1 or 2
* Mini-Mental Test Status (MMS) > 23

Exclusion Criteria:

* Mixed non-small cell and small cell tumors
* Patients with EGFR mutated tumor
* Patient with EML4-ALK translocation
* Evolutive or symptomatic metastasis of central nervous system
* Superior vena cava syndrome
* Calcemia > 2,70 mmol/L

Ages: 70 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 632 (Actual)
Dates: Start 2013-05-16 (Actual); Primary Completion 2018-08-20 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Overall survival | Up to 15 months

SECONDARY OUTCOMES:
Feasibility of treatment (number of cycles of maintenance) | 84 days on average
  Number of cycles of maintenance (median)
Progression free survival | up to 7 months
response and stabilisation duration | up to 7 months
Number of patient with at least one adverse event | up to 7 months
Treatment duration | Up to 7 months
2nd line response rate | Up to 4 months
Number of adverse events | Up to 7 months
2nd line overall survival | Up to 7 months
2nd line progression free survival | Up to 4 months

CONTACTS AND LOCATIONS:
Locations (78):
- France (78):
  - Abbeville - CH, Abbeville
  - Centre Hospitalier du Pays d'Aix, Aix-en-Provence
  - Amiens - CHU, Amiens
  - Clinique de l'Europe, Amiens
  - Annecy - CH, Annecy
  - Auxerre - CH, Auxerre
  - CH de la Côte Basque, Bayonne
  - CHU Besancon - Pneumologie, Besançon
  - Blois - CH, Blois
  - APHP - CHU Avicenne - Oncologie Medicale, Bobigny
  - CH Pierre Oudot, Bourgoin
  - Brest - Clinique Pasteur, Brest
  - Caen - Centre François Baclesse, Caen
  - CHU Côte de Nâcre, Caen
  - CH Cahors, Cahors
  - CH de Cannes, Cannes
  - Chauny - CH, Chauny
  - Hôpital de Cholet - Pneumologie, Cholet
  - Clamart - Hôpital Percy, Clamart
  - Hôpitral Gabriel Montpied - Pneumologie, Clermont-Ferrand
  - CH, Colmar
  - CH Compiègne - Pneumologie, Compiègne
  - CHI Créteil, Créteil
  - CH de Dax, Dax
  - CHU Hôpital du Bocage, Dijon
  - Foix - CH, Foix
  - CHU Grenoble - pneumologie, Grenoble
  - Saint Omer - CHI, Helfaut
  - Jonzac - CH, Jonzac
  - Chartres - CH, Le Coudray
  - Le Mans - Centre Hospitalier, Le Mans
  - Institut d'Oncologie Hartmann, Levallois-Perret
  - CH de Longjumeau, Longjumeau
  - Lorient - CHBS, Lorient
  - Lyon - Clinique Mutualiste, Lyon
  - CH Saint Joseph Saint Luc, Lyon
  - Hôpital de la Croix Rousse, Lyon
  - Hôpital Louis Pradel, Lyon
  - Lyon - Clinique de la Sauvegarde, Lyon
  - Lyon - Hôpital Jean Mermoz, Lyon
  - Hôpital Ambroise Paré, Marseille
  - Hôpital Nord - Oncologie Multidisciplinaire & Innovations Thérapeutiques, Marseille
  - Institut Paoli Calmette, Marseille
  - Maubeuge - Polyclinique du Parc, Maubeuge
  - Polyclinique du Val de Sambre, Maubeuge
  - CH de Macon, Mâcon
  - Metz - Belle Isle, Metz
  - Mont de Marsan - CH, Mont-de-Marsan
  - Montargis - CH, Montargis
  - Montbéliard - CH, Montbéliard
  - Centre Hospitalier, Montélimar
  - Montpellier - CHRU, Montpellier
  - Mulhouse - CH, Mulhouse
  - CHU Nancy, Nancy
  - Nevers - CH, Nevers
  - Centre Antoine Lacassagne, Nice
  - Orléans - CH, Orléans
  - Paris - Saint Louis, Paris
  - Hopital Tenon - Pneumologie, Paris
  - GH Paris Saint-Joseph, Paris
  - CHG de Pau, Pau
  - Perpignan - Centre Catalan d'Oncologie, Perpignan
  - Perpignan - Ch, Perpignan
  - Lyon Sud, Pierre-Bénite
  - Rennes - CHU, Rennes
  - Roubaix - CH, Roubaix
  - Saint-Nazaire - Clinique Mutualiste de l'Estuaire, Saint-Nazaire
  - Centre Hospitalier, Saint-Quentin
  - Strasbourg - NHC, Strasbourg
  - Suresnes - Hopital Foch, Suresnes
  - Toulon - CHI, Toulon
  - Hôpital Larrey - Pneumologie, Toulouse
  - Tours - CHU, Tours
  - Troyes - CH, Troyes
  - Valenciennes - Clinique, Valenciennes
  - Vernon - CHI, Vernon
  - Versailles - CH, Versailles
  - CH de Villefranche - Pneumologie, Villefranche

REFERENCES:
- [Background] Quoix E, Zalcman G, Oster JP, Westeel V, Pichon E, Lavole A, Dauba J, Debieuvre D, Souquet PJ, Bigay-Game L, Dansin E, Poudenx M, Molinier O, Vaylet F, Moro-Sibilot D, Herman D, Bennouna J, Tredaniel J, Ducolone A, Lebitasy MP, Baudrin L, Laporte S, Milleron B; Intergroupe Francophone de Cancerologie Thoracique. Carboplatin and weekly paclitaxel doublet chemotherapy compared with monotherapy in elderly patients with advanced non-small-cell lung cancer: IFCT-0501 randomised, phase 3 trial. Lancet. 2011 Sep 17;378(9796):1079-88. doi: 10.1016/S0140-6736(11)60780-0. Epub 2011 Aug 8. PMID 21831418
- [Result] Quoix E, Audigier-Valette C, Lavole A, Molinier O, Westeel V, Barlesi F, Le Treut J, Pichon E, Dauba J, Otto J, Moreau L, Madelaine J, Dumont P, Margery J, Debieuvre D, Renault PA, Pujol JL, Langlais A, Morin F, Moro-Sibilot D, Souquet PJ. Switch maintenance chemotherapy versus observation after carboplatin and weekly paclitaxel doublet chemotherapy in elderly patients with advanced non-small cell lung cancer: IFCT-1201 MODEL trial. Eur J Cancer. 2020 Oct;138:193-201. doi: 10.1016/j.ejca.2020.07.034. Epub 2020 Sep 6. PMID 32898792
- See also: IFCT official website — http://www.ifct.fr

DOCUMENTS (1):
  • Study Protocol (2015-11-20): https://cdn.clinicaltrials.gov/large-docs/03/NCT01850303/Prot_000.pdf